CLINICAL TRIAL: NCT01887171
Title: A Randomized Study of Effect of Preimplantation Portal Vein and Hepatic Artery Liver Flushing With Tacrolimus on Ischemia-reperfusion Injury, Allograft Dysfunction and Liver Histology
Brief Title: Evaluation of Preimplantation Portal Vein and Hepatic Artery Flushing With Tacrolimus
Acronym: PATAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Republican Scientific and Practical Center for Organ and Tissue Transplantation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1633
Record Dates: First submitted 2013-04-06; First posted 2013-06-26 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2014-11

CONDITIONS: Early Allograft Dysfunction; Ischemic Reperfusion Injury; Liver Transplantation; Hyperfibrinolysis
Keywords: Liver transplantation; Early allograft dysfunction; Ischemic reperfusion injury; Portal and arterial ex vivo HTK flush
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus + HTK (Experimental): During back-table operation 1000 ml of HTK solution cooled to 2-4˚C containing 20 ng/ml Tacrolimus would be given through intraportal (under gravity pressure of 40 cm H2O) and intraarterial infusion (under pressure of 40-50 mm Hg) followed by intraportal infusion of 200 ml 5% solution of Albumin containing 20 ng/ml Tacrolimus under gravity pressure of 40 cm H2O.
  Interventions: Drug: Tacrolimus
- HTK (No Intervention): During back-table operation 1000 ml of HTK solution cooled to 2-4˚C would be given through intraportal (under gravity pressure of 40 cm H2O) and intraarterial infusion (under pressure of 40-50 mm Hg) followed by intraportal infusion of 200 ml 5% solution of Albumin under gravity pressure of 40 cm H2O.

INTERVENTIONS:
Drug: Tacrolimus — 1000 ml of HTK solution (Custodiol, Dr. Franz Köhler Chemie GmBH) cooled to 2-4˚C containing 20 ng/ml Tacrolimus would be given through intraportal (under gravity pressure of 40 cm H2O) and intraarterial infusion (under pressure of 40-50 mm Hg) followed by intraportal infusion of 200 ml 5% solution of Albumin containing 20 ng/ml Tacrolimus under gravity pressure of 40 cm H2O.
  Other Names: Tacrolimus, Astellas Pharma Europe; Custodiol, Dr. Franz Köhler Chemie GmBH
  Arms: Tacrolimus + HTK

SUMMARY:
The purpose of this study is to determine whether the Tacrolimus added to histidine-tryptophan-ketoglutarate (HTK) solution given through intraportal and intraarterial infusion during back-table procedure is capable of reducing the degree of early allograft liver dysfunction, as assessed by postoperative levels of aspartate aminotransferase (AST), alanine aminotransferase (ALT), during first 7 postoperative days and by serum and histochemical markers of liver injury and inflammation.

DETAILED DESCRIPTION:
Early allograft liver dysfunction remains a significant complication of cadaveric liver transplantation with resource consuming and costly treatment, increased risk of multiorgan failure and 6-months mortality.

Ischemic reperfusion injury (IRI) is a main reason for early allograft liver dysfunction. Inflammatory response to brain death in donor can precipitate the extent of dysfunction after reperfusion in recipient (1). Clear inflammatory pathways in response to IRI have been reported to be associated with early allograft liver dysfunction (2,3). It was shown that ex vivo intraportal tacrolimus perfusion suppressed inflammation and immune response in the transplanted liver on a genome-wide basis (4).

We hypothesize that Tacrolimus added to HTK solution given through intraportal and intraarterial back-table infusion is capable of reducing the degree of early allograft liver dysfunction, as assessed by incidence of postreperfusion hyperfibrinolysis, postoperative levels of AST,ALT, during 1-7 postoperative days as well as serum and histochemical markers of liver injury and inflammation compared to no intraportal and intraarterial back-table infusion.

ELIGIBILITY:
Inclusion Criteria:

* Donor:

age 15-65 years macrovesicular steatosis < 40% (macroscopy or biopsy) sodium <165 mmol/l ICU stay and ventilation < 11 days cold ischemia time < 13 hours AST < 200 U/l ALT < 200 U/l bilirubin < 50 μmol/l application of norepinephrine is allowed

* Recipient age: 18-69

Exclusion Criteria:

Recipient:

* live donor liver transplant
* reduced and split grafts
* multi organ failure

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aliaksei E Shcherba, PhD, Principal Investigator — RSPC for tissue and organ transplantation; Oleg O Rumo, MD PhD, Study Chair — RSPC for organ and tissue transplantation, Minsk 9th clinic
Locations (1):
- RSPC for organ and tissue transplantation, Minsk 9th clinic, Minsk, Belarus

REFERENCES:
- [Background] Friedman BH, Wolf JH, Wang L, Putt ME, Shaked A, Christie JD, Hancock WW, Olthoff KM. Serum cytokine profiles associated with early allograft dysfunction in patients undergoing liver transplantation. Liver Transpl. 2012 Feb;18(2):166-76. doi: 10.1002/lt.22451. PMID 22006860
- [Background] Busuttil RW, Tanaka K. The utility of marginal donors in liver transplantation. Liver Transpl. 2003 Jul;9(7):651-63. doi: 10.1053/jlts.2003.50105. PMID 12827549
- [Background] Ilmakunnas M, Tukiainen EM, Rouhiainen A, Rauvala H, Arola J, Nordin A, Makisalo H, Hockerstedt K, Isoniemi H. High mobility group box 1 protein as a marker of hepatocellular injury in human liver transplantation. Liver Transpl. 2008 Oct;14(10):1517-25. doi: 10.1002/lt.21573. PMID 18825712
- [Background] Kristo I, Wilflingseder J, Kainz A, Marschalek J, Wekerle T, Muhlbacher F, Oberbauer R, Bodingbauer M. Effect of intraportal infusion of tacrolimus on ischaemic reperfusion injury in orthotopic liver transplantation: a randomized controlled trial. Transpl Int. 2011 Sep;24(9):912-9. doi: 10.1111/j.1432-2277.2011.01284.x. Epub 2011 Jun 14. PMID 21672049
- [Background] Olthoff KM, Kulik L, Samstein B, Kaminski M, Abecassis M, Emond J, Shaked A, Christie JD. Validation of a current definition of early allograft dysfunction in liver transplant recipients and analysis of risk factors. Liver Transpl. 2010 Aug;16(8):943-9. doi: 10.1002/lt.22091. PMID 20677285
- [Result] Shcherba A.E., Minou A.F., Efimov D.J., Korotkov S.V., LebedzO.A., Dzyadzko A.M., Karitka A., Santotski E.O., Rummo O.O.//Influence of Back Table Portal And Arterial Flushing with HTK and Tacrolimus on the Incidence of Liver Graft Dysfunction. Materials of "Avantguardia in the HPB - surgery and Liver transplantation: When East meets West". Volume 61, June 2014, Supplement 1.- P. S13-14.
- [Result] Abstracts of the ILTS 20(th) Annual International Congress, June 3-7, 2014, London, United Kingdom. Liver Transpl. 2014 Jun;20 Suppl 1:S1-399. doi: 10.1002/lt.23901. No abstract available. PMID 25044812
- See also: Related Info — http://journal.transpl.ru/vtio/article/view/561/488
- See also: Related Info — http://www.jtmr.ro/article/portal-and-arterial-flushing-with-htk-and-tacrolimus-can-attenuate-the-incidence-of-early-liver-allograft-dysfunction
- Available data/document: Clinical Study Report: 10.15825/1995-1191-2015-3-24 — http://journal.transpl.ru/vtio/article/view/561/488
- Available data/document: Clinical Study Report: 10.21614/jtmr-21-2-82 — http://www.jtmr.ro/article/portal-and-arterial-flushing-with-htk-and-tacrolimus-can-attenuate-the-incidence-of-early-liver-allograft-dysfunction

RESULTS

PARTICIPANT FLOW:
Groups:
- HTK Solution Only: During back-table operation 1000 ml of HTK solution cooled to 2-4˚C would be given through intraportal (under gravity pressure of 40 cm H2O) and intraarterial infusion (under pressure of 40-50 mm Hg) followed by intraportal infusion of 200 ml 5% solution of Albumin under gravity pressure of 40 cm H2O.
Period: Overall Study
Arm/Group | Tacrolimus + HTK | HTK Solution Only
Started | 43 | 43
Completed | 43 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- HTK Only: During back-table operation 1000 ml of HTK solution cooled to 2-4˚C would be given through intraportal (under gravity pressure of 40 cm H2O) and intraarterial infusion (under pressure of 40-50 mm Hg) followed by intraportal infusion of 200 ml 5% solution of Albumin under gravity pressure of 40 cm H2O.
- Total: Total of all reporting groups
Arm/Group | Tacrolimus + HTK | HTK Only | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 42 | 84
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 50 [38 to 56] | 50 [40 to 58] | 50 [38 to 58]
Gender [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 25 | 22 | 47
Region of Enrollment [Number; unit: participants]
  Belarus | 43 | 43 | 86

OUTCOME MEASURES:

1. Primary Outcome: Early Allograft Dysfunction
Description: Protocol is restricted to liver transplants performed with classic technique with sequential portal-arterial reperfusion.
  Early allograft dysfunction will be assessed on the basis of highest levels of AST and ALT during 1-7 postoperative days.
Time Frame: 1-7 postoperative days after liver transplant procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus + HTK | HTK Solution Only
Number analyzed (Participants) | 43 | 43
Participants | 6 | 18

2. Secondary Outcome: Ischemic Reperfusion Injury of the Liver Allograft
Description: Protocol is restricted to liver transplants performed with classic technique with sequential portal-arterial reperfusion.
  A wedge resection of small (5x5mm) part of liver segment-III will be sampled at 2 hours after venous reperfusion. Rate of necrosis, inflammation, vascular thrombosis, cluster of differentiation (CD) 68 and High mobility group box 1 protein (HMGB1) staining will be assessed thereafter.
Time Frame: liver biopsy taken at 2 hours after portal reperfusion
Reporting Status: Not Posted

3. Secondary Outcome: Inflammatory Response to Reperfusion
Description: Protocol is restricted to liver transplants performed with classic technique with sequential portal-arterial reperfusion.
  After unclamping portal vein but before unclamping the inferior vena cava and after venting of first 100 ml of blood a 5 ml sample of blood (code is "HV") from a tube inserted into caval suture line will be taken. Another 5 ml sample of blood (code is "C") will be taken by puncture of one of hepatic veins 20 min later. Samples (5 ml each) of peripheral blood will be taken on 1st and 3d postoperative day (POD). P-selectin, interleukin-6, interleukin-8, tumor necrosis factor alfa (TNF-a) and macrophage inflammatory protein 1 alpha (MIP-1a) will be determined in samples "HV" and "C". Interleukin-8, elastase, TNF-a and vascular endothelial growth factor (VEGF) will be determined in samples of 1st and 3d POD.
Time Frame: 0 and 20 min after portal reperfusion, 1 and 3 postoperative day
Reporting Status: Not Posted

4. Secondary Outcome: Postreperfusion Hyperfibrinolysis
Description: Protocol is restricted to liver transplants performed with classic technique with sequential portal-arterial reperfusion.
  Peripheral blood samples will be taken 15 min and 2 hours after portal reperfusion.
  Hyperfibrinolysis will be diagnosed by Thromboelastometry (ROTEM) if one or more following criteria are met:
  LI30<85% or ML>15% or LI60<85% or A10 in Extem is by 15% is less then A10 in Aptem.
Time Frame: 15 min and 2 hours after portal reperfusion
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- HTK Solution: During back-table operation 1000 ml of HTK solution cooled to 2-4˚C would be given through intraportal (under gravity pressure of 40 cm H2O) and intraarterial infusion (under pressure of 40-50 mm Hg) followed by intraportal infusion of 200 ml 5% solution of Albumin under gravity pressure of 40 cm H2O.
Arm/Group | Tacrolimus + HTK | HTK Solution
Serious Adverse Events (participants affected / at risk) | 8/12 | 20/22
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus + HTK (N=12) | HTK Solution (N=22)
Early allograft dysfunction (Hepatobiliary disorders) | 6 (6) | 18 (18) — defined due to Olthoff criteria (2010)
Death (Surgical and medical procedures) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No